CLINICAL TRIAL: NCT01580605
Title: Prospective, Longitudinal and National Follow-up Program of Adult Patients With Somatotropic Hormone Deficiency for Whom Substituting Treatment by Norditropin SimpleXx Was Started
Brief Title: French National Registry of Adults With Growth Hormone Deficiency Treated With Somatropin
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GHDA-1755
Record Dates: First submitted 2012-04-13; First posted 2012-04-19 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Users of somatropin
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Data are extracted from the French National Registry "l'Observatoire National des Prescriptions et Consommations de Médicaments" to where physicians report data about growth hormone treatment

SUMMARY:
This study is conducted in Europe. The aim of this study is to extract data from the French National Registry holding information about patients having initiated growth hormone therapy with the objective to describe patients receiving growth hormone therapy, assess efficacy and safety of somatropin (Norditropin® SimpleXx®) and evaluate treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adult with growth hormone deficiency
* Treated with Norditropin® SimpleXx (somatropin)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients with growth hormone deficiency and treated with Norditropin® SimpleXx (somatropin) for whom Norditropin® SimpleXx® has been initiated either before or during the registry inclusion period
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2003-07-17 (Actual); Primary Completion 2011-11-28 (Actual); Study Completion 2011-11-28 (Actual)

PRIMARY OUTCOMES:
Weight | Once a year for 5 years
Body composition | Once a year for 5 years
Waist:Hip Ratio | Once a year for 5 years
Body mass index (BMI) | Once a year for 5 years

SECONDARY OUTCOMES:
IGF-1 (Insulin-like growth factor 1) concentration | Once a year for 5 years
Lipids: Total cholesterol, high-density lipoprotein (HDL), low-density lipoprotein (LDL) and triglycerides | Once a year for 5 years
Dose prescribed | Once a year for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Lyon, France

REFERENCES:
- [Derived] Borson-Chazot F, Chabre O, Salenave S, Klein M, Brac de la Perriere A, Reznik Y, Kerlan V, Hacques E, Villette B. Adherence to growth hormone therapy guidelines in a real-world French cohort of adult patients with growth hormone deficiency. Ann Endocrinol (Paris). 2021 Feb;82(1):59-68. doi: 10.1016/j.ando.2020.11.007. Epub 2020 Dec 5. PMID 33290752
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com